CLINICAL TRIAL: NCT06981533
Title: Efficacy of Auricular Acupressure in Treating Premenstrual Syndrome in Female Undergraduate Students
Brief Title: Auricular Acupressure for Premenstrual Syndrome in Female Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Le Nguyen Thanh Vy, MD, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4259/QĐ-ĐHYD; 30.000.000 VND (Other Grant/Funding Number: University of Medicine and Pharmacy at Ho Chi Minh City)
Record Dates: First submitted 2025-05-03; First posted 2025-05-20 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Syndrome; Auricular Acupressure; Female undergraduate students; PMS; The Premenstrual Symptoms Screening Tool
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Intervention Model Description: A randomized, single-blind, parallel controlled trial
Who Masked: Participant
Masking Description: Participants: They did not know about auricular acupuncture, auricular acupressure. The investigator informs the information about the specific location of the acupoints used and the purpose of the study. The investigator provided a questionnaire to assess the participants's knowledge of auricular acupuncture, auricular acupressure, expectations, and motivation to participate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular acupressure therapy + Lifestyle modifications (Experimental): Auricular acupressure therapy once a week on one ear for a total of 8 weeks (8 sessions), with treatment alternating between the two ears.
  Lifestyle modifications were followed according to the guidelines of the Royal College of Obstetricians and Gynaecologists (RCOG 2017) on PMS management.
  Interventions: Other: Auricular acupressure therapy; Other: Lifestyle modifications
- Sham auricular acupressure therapy + Lifestyle modifications (Sham Comparator): Sham auricular acupressure once a week on one ear for a total of 8 weeks (8 sessions), with treatment alternating between the two ears.
  Lifestyle modifications were followed according to the guidelines of the Royal College of Obstetricians and Gynaecologists (RCOG 2017) on PMS management.
  Interventions: Other: Sham auricular acupressure therapy; Other: Lifestyle modifications

INTERVENTIONS:
Other: Auricular acupressure therapy — Auricular acupressure will be performed using Cowherb seeds (Wangbuliuxing seeds) applied to specific acupoints, including Shenmen (TF4), Sympathetic (AH6a), Endocrine (CO18), Liver (CO12), Kidney (CO10), Subcortex (AT4), and Zero Point on one ear, with treatment administered once a week, alternating between the left and right ears. In total, auricular acupressure was applied 8 times over a period of 8 weeks. The first treatment session occurred 5-7 days prior to the onset of menstruation. Participants were instructed to perform acupressure at the acupoint sites three times daily-morning, noon, and evening-pressing each point for 1 minute per session.
  Other Names: Auricular Acupressure; Ear Acupressure
  Arms: Auricular acupressure therapy + Lifestyle modifications
Other: Sham auricular acupressure therapy — Sham auricular acupressure therapy will be performed using similarly sized adhesive patches without seeds, applied to the same acupoint locations as in the intervention group. The procedure steps and the duration of the trial were the same as in the auricular acupressure group.
  Other Names: Sham Ear Acupressure
  Arms: Sham auricular acupressure therapy + Lifestyle modifications
Other: Lifestyle modifications — Lifestyle modifications will be followed according to the "Guidelines for the Management of Premenstrual Syndrome" by the Royal College of Obstetricians and Gynaecologists (RCOG), which will include: Regular moderate exercise (such as walking, yoga, or swimming), stress reduction, and ensuring quality sleep (7-8 hours per night); Reducing intake of salt, sugar, and foods containing saturated fats; Increasing intake of high-fiber foods such as fruits and vegetables; Avoiding smoking, and limiting alcohol, and other stimulants.
  Other Names: Lifestyle changes

SUMMARY:
Premenstrual Syndrome (PMS) is a common gynecological disorder that significantly affects the quality of life for women of reproductive age, with symptoms including emotional, behavioral, and physical disturbances occurring approximately one week before menstruation. PMS is especially prevalent among female undergraduate students, who often experience heightened stress due to academic pressures and lack emotional coping strategies. While pharmacological treatments, such as SSRIs and hormonal therapies, have been used to manage PMS symptoms, they may have side effects and are not always effective in the long term. This has led to increasing interest in alternative treatments such as traditional medicine. Auricular acupressure, a non-invasive and low-risk method, has shown promising results in managing PMS symptoms and is gaining attention as a possible solution.

The goal of this clinical trial is to evaluate the efficacy and safety of auricular acupressure in reducing PMS symptoms in female undergraduate students. The main questions it aims to answer are:

* Does auricular acupressure reduce the severity of PMS symptoms in female undergraduate students?
* Is auricular acupressure safe and well-tolerated by participants? Researchers will compare the intervention group (receiving auricular acupressure) to the control group (receiving sham auricular acupressure) to see if auricular acupressure has a significant impact on reducing PMS symptoms and improving quality of life.

Participants will:

* Receive auricular acupressure on specific acupoints or sham treatment.
* Complete assessments of PMS symptoms using the Premenstrual Symptoms Screening Tool (PSST) at baseline, 1 week, and 8 weeks.
* Complete a quality of life assessment using the WHOQOL-Bref scale at the same time points.
* Be monitored for any adverse effects during the 8-week trial period.

DETAILED DESCRIPTION:
Participants and Methods: A randomized, single-blind, controlled trial was conducted with 60 female undergraduate students, aged 18 to 25 years, residing in Ho Chi Minh City, who exhibit symptoms of Premenstrual Syndrome (PMS) were eligible for inclusion. Participants were required to meet the inclusion criteria and not fall under any exclusion criteria.

Participants were randomly assigned into two groups in a 1:1 ratio: the intervention group received auricular acupressure using Cowherb seeds (Wangbuliuxing seeds) applied to specific acupoints, including Shenmen (TF4), Sympathetic (AH6a), Endocrine (CO18), Liver (CO12), Kidney (CO10), Subcortex (AT4), and Zero Point, while the control group received a sham treatment. The sham treatment involved a patch of similar size to the Cowherb seed patch but without any active ingredients, applied to the same acupoint locations as the intervention group.

Both groups were provided with instructions on lifestyle changes to help manage PMS symptoms. The intervention lasted for 8 weeks (2 menstrual cycles), with weekly patch changes alternating between the left and right ears. PMS symptoms were assessed using the Premenstrual Symptoms Screening Tool (PSST), and quality of life was measured using the WHOQOL-Bref scale. Data were collected at baseline, after 1 week, and after 8 weeks. Adverse effects were carefully monitored throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Female students aged 18 to 25 with active menstrual cycles and menstrual periods ranging from 25 to 35 days.
* Participants must be able to accurately recall the start date of their most recent menstruation cycle.
* Participants must exhibit symptoms of Premenstrual Syndrome (PMS) and meet the diagnostic criteria for PMS as defined by the American College of Obstetricians and Gynecologists (ACOG) 2014.
* Participants must not have any chronic conditions, including respiratory diseases (e.g., asthma, pneumonia, chronic obstructive pulmonary disease), thyroid disorders, autonomic nervous system disorders, hypertension, coronary artery disease, or diabetes, as determined through clinical examination, medical history, and prior medical records.
* Participants must not have severe psychological stress (a score lower than 27 on the Perceived Stress Scale - PSS-10).
* Participants must be mentally alert and in good contact with the researcher.
* Participants must voluntarily consent to participate in the study.
* Participants must not have prior knowledge of auricular acupuncture or auricular acupressure.

Exclusion Criteria:

* Infection or lesions in the ear area (e.g., scars, tears, abrasions).
* Menstrual cycles shorter than 25 days or longer than 35 days.
* Participants unable to recall the start date of their most recent menstruation cycle.
* Participants diagnosed with gynecological conditions such as uterine fibroids, endometriosis, or ovarian cysts, based on medical history and recent abdominal ultrasound results (within the past 6 months).
* History of abortion, currently pregnant, or planning to become pregnant during the study period.
* Use of antidepressants and/or antipsychotic drugs, hormone supplements, oral contraceptives, or intrauterine devices within the past two months.
* Current or past psychiatric disorders.
* Participants with severe psychological stress (a score between 27 and 40 on the PSS-10).
* Unstable mental state, sensory impairments (e.g., hearing, vision, speech), or cognitive disabilities.
* Previous auricular acupressure, acupuncture, or other forms of acupuncture for PMS treatment within the last 6 months.
* Use of medication for PMS symptom relief during the study period.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
The change in PSST scores | From baseline to 1 week and to the end of treatment at 8 weeks
  This is a quantitative variable, with the unit being score. Scoring is done by asking participants based on the Premenstrual Symptoms Screening Tool (PSST) with 19 items. Each item is scored according to the Likert-4 scale, and the total score from the 19 items represents the overall PMS symptom score.
The change in WHOQOL-Bref scores | From baseline to 1 week and to the end of treatment at 8 weeks
  This is a quantitative variable, with the unit being points. The scoring is done by asking participants 26 questions to assess various domains of quality of life, including Physical Health, Psychological, Social Relationships, and Environment. Responses are categorized based on the Likert-5 scale. The average score for each domain is converted to a 100-point scale.

SECONDARY OUTCOMES:
Adverse effects | Through study completion, an average of 8 weeks
  Adverse effects occurring during the treatment and follow-up periods, regardless of their association with the interventions, will be recorded and managed with appropriate measures.

CONTACTS AND LOCATIONS:
Overall Officials: Deputy principal, Study Chair — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- Faculty of Traditional medicine - University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Korelo RIG, Moreira NB, Miguel BAC, Cruz CGD, Souza NSP, Macedo RMB, Gallo RBS. Effects of Auriculotherapy on treatment of women with premenstrual syndrome symptoms: A randomized, placebo-controlled clinical trial. Complement Ther Med. 2022 Jun;66:102816. doi: 10.1016/j.ctim.2022.102816. Epub 2022 Feb 12. PMID 35167949
- [Background] Koleini S, Valiani M. Comparing the Effect of Auriculotherapy and Vitamin B6 on the Symptoms of Premenstrual Syndrome among the Students who Lived in the Dorm of Isfahan University of Medical Sciences. Iran J Nurs Midwifery Res. 2017 Sep-Oct;22(5):354-358. doi: 10.4103/ijnmr.IJNMR_120_16. PMID 29033988
- [Background] Jang SH, Kim DI, Choi MS. Effects and treatment methods of acupuncture and herbal medicine for premenstrual syndrome/premenstrual dysphoric disorder: systematic review. BMC Complement Altern Med. 2014 Jan 10;14:11. doi: 10.1186/1472-6882-14-11. PMID 24410911
- [Background] Zhang J, Cao L, Wang Y, Jin Y, Xiao X, Zhang Q. Acupuncture for Premenstrual Syndrome at Different Intervention Time: A Systemic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2019 Jun 25;2019:6246285. doi: 10.1155/2019/6246285. eCollection 2019. PMID 31341497
- [Background] Armour M, Ee CC, Hao J, Wilson TM, Yao SS, Smith CA. Acupuncture and acupressure for premenstrual syndrome. Cochrane Database Syst Rev. 2018 Aug 14;8(8):CD005290. doi: 10.1002/14651858.CD005290.pub2. PMID 30105749